CLINICAL TRIAL: NCT06561529
Title: A Prospective, Open-label, Single-arm Clinical Study to Evaluate the Safety and Performance of the Gastric Bypass Stent System as a Treatment for Hepatic Fibrosis in Obese Patients in European Region
Brief Title: The Gastric Bypass Stent System as a Treatment for Hepatic Fibrosis in Obese Patients in European Region
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MDCECRO LLC (Network)
Collaborators: Hangzhou Tangji Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-LV01-001
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Fibrosis; Liver
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group, subjects will be treated with the Gastric Bypass Stent System implanted (Experimental): In total, 10 subjects will be enrolled from 2 investigational sites located in Latvia. Any subject participating in this clinical investigation will not be replaced once withdrawn or lost to follow-up. This study includes 3 phases; screening period, procedural period, and a follow-up period. Following screening, subjects will be treated with the Gastric Bypass Stent System implanted under gastroscopy (Visit 3; Day 0).
  Interventions: Device: Gastric Bypass Stent System

INTERVENTIONS:
Device: Gastric Bypass Stent System — The Gastric Bypass Stent System is intended to be used in weight loss treatment for obesity holds potential as a non-invasive technique for managing hepatic fibrosis. This clinical investigation will be used to evaluate the safety and performance of the investigational device for the intended use.

SUMMARY:
The Gastric Bypass Stent System is intended to be used in weight loss treatment for obesity and holds potential as a non-invasive technique for managing hepatic fibrosis. This pilot, prospective, single-arm, clinical investigation aims to evaluate the safety and performance of the Gastric Bypass Stent System for hepatic fibrosis treatment in Europe. This clinical investigation and the ongoing clinical investigation (Protocol number: BL-RD08-040) will be used to evaluate the safety and performance of the investigational device for the intended use.

ELIGIBILITY:
Subjects who meet all of the following criteria are eligible for this clinical investigation:

1. Age 18-65 years.
2. BMI ≥ 30 kg/m².
3. Medical history suggests suspected or confirmed NASH fibrosis. Meeting any of the following criteria indicates NASH liver fibrosis:

   * Historical biochemical tests for fibrosis: PRO-C3 >14 ng/mL or ELF ≥9
   * Fibroscan, transient elastography ≥8.5 kPa, controlled attenuation parameter ≥280 dB/m
   * Based on existing pathology review, liver biopsy within <2 years before the expected randomization shows stage 1B, 2, or 3 fibrosis NASH, with no significant weight change >5% or medications likely affecting NAS or fibrosis stage.
4. Liver biopsy confirming NASH within 6 months before the randomization date, with liver biopsy fibrosis stage 1-3, NAS ≥3, and at least a score of 1 for the following NAS components:

   * Steatosis (0-3 points)
   * Ballooning (0-2 points)
   * Lobular inflammation (0-3 points)
5. Patients who have not achieved effective results after three months of lifestyle modifications and non-invasive treatments (non-diabetic patients have not achieved a weight loss of 5%, diabetic patients have not achieved a weight loss of 3%).
6. Able and willing to provide informed consent for participation in the clinical investigation and comply with all study procedures and assessments.

Subjects who meet any of the following criteria are not eligible for this clinical investigation:

1. Patients with liver cirrhosis
2. Patients with secondary obesity; a medical condition that has caused weight gain such as endocrine disorders and hypothalamic disorders.
3. Chronic, daily use of systemic anti-inflammatory or corticosteroid medications (e.g., ibuprofen, prednisolone) for more than 1 week (not including low-dose aspirin for cardiac prophylaxis or inhaled corticosteroids).
4. Patients with less than one-year continuous treatment before baseline with hypoglycemic drugs with known weight loss effects (e.g., GLP-1 agonists, SGLT-2 inhibitors, DDP-4 inhibitors).
5. Patients diagnosed with type 1 diabetes.
6. Patients with the function of islet β cell basically lost, C-peptide ≤ 1/2 of the normal low limit, or low and flat C-peptide release curve under glucose load.
7. Patients with significant iron deficiency or iron deficiency anemia upon the Investigator's discretion.
8. Patients with coagulation dysfunction and chronic, daily use of systemic anti-inflammatory or anti-coagulation medication in the past month (not including low-dose aspirin).
9. Patients with severe liver and kidney dysfunction, and a serum creatinine concentration ≥ 180 μmol/L.
10. Patients with Class III heart function of New York Heart Association Functional Classification (NYHA) or higher upon the Investigators evaluation.
11. Patients who have undergone Endoscopic Retrograde Cholangiopancreatography (ERCP) or have a history of cholecystitis or liver abscess, as assessed by medical history and abdominal ultrasound.
12. Patients with a duodenal ulcer, gastric ulcer, or previous and existing pancreatitis, as assessed by abdominal ultrasound, gastroscopy (prior to the procedure at Visit 3), and medical history.
13. Patients with gallstones (diameter ≥ 20 mm) with clinical symptoms as assessed by abdominal ultrasound and medical history.
14. Patients with on-going thyroid dysfunction, not stabilized despite appropriate treatment.
15. Patients with hemorrhage or potential hemorrhage in the digestive tract.
16. Patients with gastrointestinal tract anomalies, such as gastrointestinal tract atresia, or other conditions that would result in failed placement in the gastrointestinal tract, as assessed by gastroscopy (prior to the procedure at Visit 3), abdominal digital gastrointestinal radiography, and medical history.
17. Patients with a history of bowel obstruction or related diseases in the past year.
18. Patients with a history of systemic lupus erythematosus or scleroderma.
19. Patients with severe infections that are not controlled.
20. Patients with poor general condition and having endoscopic contraindications (as evaluated by the Investigator).
21. Pregnant women or planning to become pregnant.
22. Patients with an alcohol dependence or substance abuse.
23. Patients with unstable psychiatric disorders.
24. Patients who are enrolled in another investigational study and have not completed the required follow-up period.
25. Patients with an allergy to any of the components of the investigational device.
26. Patients with any other conditions evaluated by the Investigators as unsuitable for participating in the clinical investigation.
27. Patients who are positive for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus as determined by antibodies, deoxy/ribonucleic acid (DNA/RNA), or antigens.

Note: Anti-HCV positive, but HCV-RNA negative HCV patients can be included, based on investigator's judgement, if it's not the primary reason for the fibrosis. Anti-HBc positive, but HBs-Ag negative patients can be included, based on investigator's judgement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Nonalcoholic Steatohepatitis Clinical Research Network (NASH CRN score) at 6 months after procedure (i.e. device implantation) | 6 months
  * Percentage of NAFLD activity score (NAS) reduction without worsening of fibrosis stage;
  * Percentage of improvement in fibrosis stage and no deterioration in NAFLD activity score (NAS)

SECONDARY OUTCOMES:
Relative percentage change in Total Weight Loss (TWL%) and changes in BMI | 12 months
  Relative percentage change in Total Weight Loss (TWL%) and changes in BMI at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.
Changes in Fibroscan Controlled Attenuation Parameter (CAP) and Liver Stiffness Measurement (LSM) | 12 months
  Changes in Fibroscan Controlled Attenuation Parameter (CAP) and Liver Stiffness Measurement (LSM) at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.
Changes in liver inflammation/injury-related markers (ALT, AST, GGT, ALP, Total Bilirubin, Direct Bilirubin) | 12 months
  Changes in liver inflammation/injury-related markers (ALT, AST, GGT, ALP, Total Bilirubin, Direct Bilirubin) at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.
Changes in blood glucose-related markers (fasting insulin, fasting glucose, fasting C-peptide) | 12 months
  Changes in blood glucose-related markers (fasting insulin, fasting glucose, fasting C-peptide, insulin resistance (HOMA-IR)) at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.
Changes in blood lipid-related markers (total cholesterol [TC], triglyceride [TG], high-density lipoprotein C [HDL-C], low-density lipoprotein C [LDL-C]), apolipoprotein A1, apolipoprotein B, apolipoprotein CIII, lipoprotein(a)) | 12 months
  Changes in blood lipid-related markers (total cholesterol [TC], triglyceride [TG], high-density lipoprotein C [HDL-C], low-density lipoprotein C [LDL-C]), apolipoprotein A1, apolipoprotein B, apolipoprotein CIII, lipoprotein(a)) at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.
Changes in blood glucose-related markers (insulin resistance (HOMA-IR)) | 12 months
  Changes in blood glucose-related markers (insulin resistance (HOMA-IR)) at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.
Changes in liver fibrosis-related markers (Forns Index) | 12 months
  Changes in liver fibrosis-related markers (Forns Index) at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.
Changes in liver fibrosis-related markers (Fibrosis-4 Index (FIB-4)) | 12 months
  Changes in liver fibrosis-related markers (Fibrosis-4 Index (FIB-4)) at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.
Changes in liver fibrosis-related markers (S Index) | 12 months
  Changes in liver fibrosis-related markers (S Index) at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.
Changes in liver fibrosis-related markers (AST to Platelet Ratio Index (APRI)) | 12 months
  Changes in liver fibrosis-related markers (AST to Platelet Ratio Index (APRI)) at 12 weeks after device implantation, at the time of device removal, 12 weeks after device removal, and 24 weeks after device removal.

CONTACTS AND LOCATIONS:
Locations (2):
- Latvia (2):
  - REUH, hospital "lnfectology center of Latvia", Riga, Rīga
  - Digestive Diseases Centre "GASTRO", Riga

IPD SHARING:
Plan to Share IPD: No